CLINICAL TRIAL: NCT05815628
Title: Next-Generation-Sequencing Approach to Neutropenic Sepsis
Acronym: NEXUS
Status: Recruiting | Type: Observational
Sponsor: Boris Böll (Other)
Collaborators: Noscendo GmbH (Unknown)
Responsible Party: Sponsor-Investigator, Boris Böll, Principal Investigator, Clinical Professor, University Hospital of Cologne
Organization: University Hospital of Cologne (Other)
Other Study IDs: NEXUS-5058
Record Dates: First submitted 2023-03-09; First posted 2023-04-18 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Febrile Neutropenia
MeSH Terms: conditions — Febrile Neutropenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: DISQVER — NGS based infection diagnosis

SUMMARY:
The aim of this prospective, observational, non-interventional, multi-centre study of the diagnostic use of DISQVER in neutropenic patients with FN is to provide further evidence of the efficacy of an NGS-based approach for detecting bloodstream infection in neutropenic patients.

DETAILED DESCRIPTION:
The aim of this prospective, observational, non-interventional, multi-centre study of the diagnostic use of DISQVER (Platform for digital pathogen diagnostics from Noscendo GmbH) in neutropenic patients with FN (Febrile neutropenia) is to provide further evidence of the efficacy of an NGS (Next-generation seqzencing)-based approach for detecting bloodstream infection in neutropenic patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Informed consent
* Neutropenia defined as <500 ANC (Absolute neutrophil Count)/µl or <1000 WBC (White bloddcell Count)/µl if ANC is not available
* Fever (with an onset < 24h) or Sepsis (with an onset <24h) Patients with a life-threatening - organ dysfunction caused by a dysregulated host response to a suspected or proven infection.

Exclusion Criteria:

* Age < 18 years
* Refusal or inability to give consent Inability to give informed consent if no acceptable patient representative is available
* Patients who had previously been included, but develop a new episode of fever during the same hospitalization, will not be included a second time
* Death is deemed imminent and inevitable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 400 neutropenic patients with febrile neutropenia
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the performance of a NGS-based | Baseline
  Number of Participants with detection of pathogen

SECONDARY OUTCOMES:
Average process time for NGS-based measurements | Baseline
  Timeframe of sampling to result of NGS-based sampling

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (6):
  - University Hospital of Cologne, Cologne
  - Hospital Dessau, Dessau
  - University Hospital of Essen, Essen
  - University Hospital of Frankfurt, Frankfurt am Main
  - University Hospital of Leipzig, Leipzig
  - University Hospital of Magdeburg, Magdeburg